CLINICAL TRIAL: NCT07013409
Title: Modulatory Effects of L. Rhamnosus LRa05 and L. Reuteri LR08 Probiotics on Hormone Metabolism, Body Composition, and Mood in Obese Women
Brief Title: Probiotics' Effects on Hormones, Body and Mood in Obese Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wecare Probiotics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: WK20250603
Record Dates: First submitted 2025-06-02; First posted 2025-06-10 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-06

CONDITIONS: Obesity, Women
MeSH Terms: conditions — Obesity | interventions — Probiotics; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic Group (Experimental): Take 30 billion CFU of complex probiotics every day (Lacticaseibacillus rhamnosus LRa05: Limosilactobacillus reuteri LR08= 1:1).
  Interventions: Dietary Supplement: Probiotic
- Placebo Group (Placebo Comparator): Taking maltodextrin 3 g/day.
  Interventions: Dietary Supplement: Maltodextrin

INTERVENTIONS:
Dietary Supplement: Probiotic — The trial period of this study is 3 months, and each patient will undergo 4 visits (in month 0, month 1, month 2, and month 3).
  Arms: Probiotic Group
Dietary Supplement: Maltodextrin — The trial period of this study is 3 months, and each patient will undergo 4 visits (in month 0, month 1, month 2, and month 3).
  Arms: Placebo Group

SUMMARY:
To evaluate the regulatory effect of probiotics formula on visceral fat metabolism and sex hormone balance in obese women.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18 to 40 years old, female, BMI ≥ 25 kg/m2.
* Be willing to receive follow-up during the intervention period.
* Be willing to provide two blood, urine and fecal samples during the intervention period.
* Be willing to take the compound probiotics by oneself every day during the intervention period.
* Have good hearing and be able to hear and understand all instructions during the intervention period.

Exclusion Criteria:

* Suffering from digestive system diseases, mainly gastrointestinal diseases (celiac disease, ulcerative colitis, Crohn's disease).
* Suffering from severe neurological disorders (epilepsy, stroke, severe head trauma, meningitis within the past 10 years, brain surgery, brain tumor, long-term coma - excluding general anesthesia).
* Have received/are currently receiving treatment for the following mental illnesses: alcohol/drug/substance abuse dependence, schizophrenia, psychosis, bipolar disorder.
* Take medication for depression or low mood.
* Suffering from internal organ failure (such as heart, liver or kidney failure, etc.).
* Have received radiotherapy or chemotherapy in the past.
* Have received general anesthesia surgery/procedures within the past three years, or plan to receive general anesthesia procedures/surgeries within the next three months during this trial.
* Have suffered from hepatitis (hepatitis B, hepatitis C), HIV or syphilis in the past.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-12-10 (Estimated)

PRIMARY OUTCOMES:
The changes of estradiol before and after the intervention | 0, 1, 2, 3 months
  The serum estrogen content of the subjects before and after the intervention was detected by enzyme-linked immunosorbent assay.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China